CLINICAL TRIAL: NCT01432379
Title: BOTOX® Prophylaxis in Patients With Chronic Migraine
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 191622-110
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- botulinum toxin Type A: 155-195 U of botulinum toxin Type A administered intramuscularly in the face, head, and neck areas as directed by physician (approximately every 12 weeks) for 1 year.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — 155-195 U of botulinum toxin Type A administered intramuscularly in the face, head, and neck areas as directed by physician (approximately every 12 weeks) for 1 year.
  Other Names: BOTOX®

SUMMARY:
This is a post authorization observational study to monitor the utilization practices and describe the safety profile of BOTOX® in clinical practice for the prophylactic treatment of headaches in adult patients with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic migraine
* Willing to use BOTOX® as preventative treatment for migraine

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Migraine
Sampling Method: Non-Probability Sample
Enrollment: 1168 (Actual)
Dates: Start 2011-09-09 (Actual); Primary Completion 2015-05-12 (Actual); Study Completion 2015-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Munich, Germany
- Oviedo, Spain
- Stockholm, Sweden
- London, United Kingdom

REFERENCES:
- [Background] Matharu M, Pascual J, Nilsson Remahl I, Straube A, Lum A, Davar G, Odom D, Bennett L, Proctor C, Gutierrez L, Andrews E, Johannes C. Utilization and safety of onabotulinumtoxinA for the prophylactic treatment of chronic migraine from an observational study in Europe. Cephalalgia. 2017 Dec;37(14):1384-1397. doi: 10.1177/0333102417724150. Epub 2017 Jul 31. PMID 28758415

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A
Started | 1168
Completed | 783
Not Completed | 385

BASELINE CHARACTERISTICS:
Population: The Treated Population includes all patients who received at least 1 dose of botulinum toxin Type A and is used for baseline characteristics.
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 1160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 977
  Male | 183

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Dysphagia
Description: Incidence rates are reported for subjects with events per 1,000 person-months and are based on the first reported occurrence of dysphagia from study enrollment up to 64 weeks. Dysphagia is difficulty or discomfort swallowing.
Time Frame: 64 weeks
Population: Treated Population: all patients who received at least 1 dose of botulinum toxin Type A
Measure: Number (95% Confidence Interval); unit: events per 1,000 person-months
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 1160
events per 1,000 person-months | 0.4 [0.1 to 0.9]

2. Secondary Outcome: Incidence Rate of Intractable Migraine
Description: Incidence rates are reported for subjects with events per 1,000 person-months and are based on the first reported occurrence of intractable migraine from study enrollment up to 64 weeks. Intractable migraine is a migraine that does not seem to go away.
Time Frame: 64 weeks
Population: Treated Population: all patients who received at least 1 dose of botulinum toxin Type A
Measure: Number (95% Confidence Interval); unit: events per 1,000 person-months
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 1160
events per 1,000 person-months | 1.6 [0.9 to 2.4]

ADVERSE EVENTS:
Description: The Treated Population includes all patients who received at least 1 dose of botulinum toxin Type A and is used to assess adverse events and serious adverse events.
Arm/Group | Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 61/1160
Other Adverse Events (participants affected / at risk) | 106/1160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=1160)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Device malfunction (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Chronic sinusitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Migraine (Nervous system disorders) | 11
Headache (Nervous system disorders) | 3
Intracranial pressure increased (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Hemiplegic migraine (Nervous system disorders) | 1
Migraine with aura (Nervous system disorders) | 1
Monoparesis (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 3
Bipolar disorder (Psychiatric disorders) | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Urge incontinence (Renal and urinary disorders) | 1
Breast haematoma (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=1160)
Migraine (Nervous system disorders) | 106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.